CLINICAL TRIAL: NCT03264339
Title: The Small Step Program - Early Intervention for Children With High Risk of Developing Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Olavs Hospital (Other)
Collaborators: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016/1366
Record Dates: First submitted 2017-08-22; First posted 2017-08-29 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Cerebral Palsy
Keywords: Infant; Hand/Growth & Development; Motor activity; Exercise; Communication
MeSH Terms: conditions — Cerebral Palsy; Motor Activity; Communication

STUDY DESIGN:
Intervention Model Description: Single-subject research design (SSRD) will be used with each participant serving as his/her own control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Smal step (Experimental): Small Step Program, comprising 3 treatment focus areas (Hand use, Mobility, Communication)
  Interventions: Behavioral: Small Step Program

INTERVENTIONS:
Behavioral: Small Step Program — The Small Step intervention program has three alternating treatment foci (Hand use, Mobility, Communication) divided into five different steps, each lasting for 6 weeks (in total 30 weeks).

SUMMARY:
Children with cerebral palsy (CP) have life-long motor disorders caused by brain injuries which occur around birth. These children go through extensive treatment during childhood, but the treatment has generally been started late due to late diagnosis (median age 15 months). New recommendations state that the clinical diagnosis "high risk of CP" should be given before 6 months corrected age, in order to be able to intervene as early as possible, and have the best possibilities to prevent or limit the adverse neurodevelopmental consequences of brain injuries occurring around birth. Thus, there is a great need to develop evidence-based early interventions for children at high risk of developing cerebral palsy.

The Small Step program is developed at Karolinska Institutet (KI) in Stockholm, Sweden and is based upon theories of brain plasticity induced by early learning. The efficacy of the program is presently being investigated at KI. Preliminary results indicate a large individual variation in response to the program among the participating children.

The aim of the present study is therefore to explore individual responses to the Small Step Program in infants at risk of developing cerebral palsy.

The main hypothesis is that infant characteristics, such as severity of brain pathology, are associated with differential response to the program. Also, infants with absent fidgety movements and children with sporadic fidgety movements are believed to respond differently to the program.

DETAILED DESCRIPTION:
The efficacy of the Small Step program is presently being investigated through a randomized controlled trial (NCT02166801) at Karolinska Institutet (KI) in Stockholm, Sweden. In the original project proposal for the current study, the plan was to contribute with inclusion of children from St. Olavs Hospital to the randomized controlled study initiated at KI. This project proposal has previously been approved by the Regional Ethical Committee (REK) for Medical Research in Mid-Norway (2016/1366). However, the researchers at KI have now completed the inclusion of participants for the randomized controlled study, and their preliminary results indicate that there is a large individual variation among the included participants regarding effect of the Small Step program. In agreement with the researchers at KI, it was therefore decided to change the design of the current study using Single Subject Research Design, a study design that is more appropriate to investigate individual response to treatment. The change in study design has been approved by REK (2016/1366-10).

Participation in this study is based on informed consent from the parents, and the child and the family participating in the project will be offered a potentially effective early intervention program that they would otherwise not be able to access.

The Small Step intervention program has three alternating treatment foci (B, C, and D) divided into five different steps, each lasting for 6 weeks (in total 30 weeks). The three treatment foci are Communication, Hand function and Mobility/gross motor function. The Hand function and Mobility steps will be conducted during two time-periods and the order will be randomised. Communication will have one intervention period during step III. The training will be conducted in the children's home by the parents on a daily basis under weekly supervision by the therapist responsible for each specific step of the intervention. General principles for the small step program are: a) collaborative goal-setting; b) promote infant's self-initiated actions; c) use of enriched home environment, d) intensity and repetition.

Before and after the intervention, there is a baseline phase with no treatment (A) and a withdrawal phase with no treatment (A), resulting in the following design: A-B-C-D-B-C-A. In addition, there is a follow-up phase when the children are 2 years of age.

ELIGIBILITY:
Inclusion Criteria:

* increased perinatal risk factors, such as preterm birth, hypoxic ischemic encephalopathy (asphyxia), and morphological brain abnormalities. These "at-risk" children are included in the regular clinical follow-up program at St. Olavs University Hospital comprising a standard examination at 3 months of age (for preterm born children: 3 months post term, so-called corrected age). At this examination, infants who exhibit two or more of the following additional risk factors will be eligible for study participation:

  * Neurological signs assessed with Hammersmith Infant Neurological Examination (HINE) with a cut-off score of < 57 (20).
  * Delayed psycho-motor development measured with Alberta Infant Motor Scale (AIMS) using 2SD as the cut-off.
  * Absent or sporadic fidgety movements assessed with the General Movements Assessment (GMA)
  * Pathological findings on cerebral imaging (magnetic resonance imaging-MRI/cerebral ultrasound) done in regular clinical practice.

Exclusion Criteria:

* unstable medical condition
* progressive disorders
* diagnosis with a specific syndrome.
* neither parent is fluent in Norwegian or English. Satisfactory skills in either language are required for participation in data collection and the coaching and education program.

Ages: 3 Months to 8 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Actual)
Dates: Start 2017-09-07 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2021-06-07 (Actual)

PRIMARY OUTCOMES:
Peabody Developmental Motor Scales, second edition (PDMS-2) | up to 2 years
  PDMS-2 is a standard measurement that assesses gross and fine motor skills in young children from birth through age 5 years. The PDMS-2 is composed of six subtests that assess related motor abilities that develop early in life. In this study, the Stationary, Locomotion, Grasping, and Visual-Motor Integration subtests will be used. The scores on these subtests are presented as percentiles, standard scores, and age equivalents.

SECONDARY OUTCOMES:
Hand Assessment for Infants (HAI) | up to 2 years
  identifies and measures upper limb asymmetry and general manual development from 3-12 months
Alberta Infant Motor Scale (AIMS) | up to 2 years
  identifies infants with delayed or deviant motor development up to 18 months of age
Gross Motor Function Measure (GMFM-66) | up to 2 years
  an observational, standardized and criterion-referenced measure, developed to evaluate change in gross motor function in children with cerebral palsy (CP)
Parent-Child Early Relational Assessment (PC-ERA) | up to 2 years
  assesses parent-child interactions to capture the affective and behavioral characteristics that parent and child bring to the interaction, and the quality or tone of the relationship
Treatment Expectancy and Credibility Survey (TCS) - modification | up to 2 years
  assesses treatment expectations

OTHER OUTCOMES:
Hammersmith Infant Neurological Examination (HINE) | at baseline, after the intervention at 30 weeks and at follow-up up at 2 years
  Identifies neurological signs in infants and is used to estimate the neurological development of infants aged two-24 months
The Working Model of the Child Interview (WMCI) | at baseline, after the intervention at 30 weeks and at follow-up up at 2 years
  a semi-structured, open-ended interview designed to assess parent´s representations of their infant/ child and their relationship with their infant/ child. The WMCI will be used to measure change over time
The Ages & Stages Questionnaire: Social and Emotional (ASQ:SE) | at baseline, after the intervention at 30 weeks and at follow-up up at 2 years
  a questionnaire to be completed by parents for assessing social and emotional difficulties in babies and young children
Norwegian Parenting Stress Index (PSI) | at baseline, after the intervention at 30 weeks and at follow-up up at 2 years
  used to measure changes in perceived parental stress over time
The Hospital Anxiety and Depression Scale (HADS) | at baseline, after the intervention at 30 weeks and at follow-up up at 2 years
  a self-assessment scale for parents and is used to detect changes in states of depression, anxiety and emotional distress over time among parents
Pediatric Evaluation of the Disability Inventory (PEDI) | at 2 years
  used to evaluate functional skills and caregiver assistance in the domains self-care, mobility, and social function over time. The child is assessed by structured interviews with the parents. The summary scores can be converted to normative standard scores and scaled scores, meaning that the child's performance will be compared with norms taken from typically developing children
Bayley Scales of Infant Development (BSID-III) | at 2 years
  a standard measurements to assess the motor (fine and gross), language (receptive and expressive), and cognitive development of infants and toddlers, ages 0-3. These scores will be used to determine the child's performance at two years of age compared with norms taken from typically developing children
Norwegian Communicative Development Inventory (NCDI) | at 2 years
  a parent questionnaire for assessing early language development of children. The NCDI involve questions about communication and language capacities corresponding to the child's ability to comprehend and use communication and language and will be collected
Structural magnetic resonance imaging (MRI)/cerebral ultrasound | before 2 years corrected age
  used to identify neuroanatomical abnormalities and underlying brain lesions. Neuroimaging data will be assessed by experienced neuroradiologists in accordance with well-established clinical assessment protocols at the hospital. This means that the children included in the project will not undergo any extra structural MRI examinations outside the normal clinical routine.
General Movements Assessment (GMA) | at 3 months corrected age
  identifies reduced movement quality (i.e. absent or sporadic fidgety movements) in infants at 3 months corrected age. The GMA is part of the clinical assessment performed at the hospital and is assessed by certified and experienced physiotherapists

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Selvaag, md, Study Director — St Olavs Hospital, Children's Clinic
Locations (1):
- St Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Yes
(in progress)

REFERENCES:
- [Background] Eliasson AC, Holmstrom L, Aarne P, Nakeva von Mentzer C, Weiland AL, Sjostrand L, Forssberg H, Tedroff K, Lowing K. Efficacy of the small step program in a randomised controlled trial for infants below age 12 months with clinical signs of CP; a study protocol. BMC Pediatr. 2016 Nov 3;16(1):175. doi: 10.1186/s12887-016-0711-x. PMID 27809886
- [Derived] Elvrum AG, Karstad SB, Hansen G, Bjorkoy IR, Lydersen S, Grunewaldt KH, Eliasson AC. The Small Step Early Intervention Program for Infants at High Risk of Cerebral Palsy: A Single-Subject Research Design Study. J Clin Med. 2024 Sep 6;13(17):5287. doi: 10.3390/jcm13175287. PMID 39274500
- [Derived] Karstad SB, Bjorseth A, Lindstedt J, Brenne AS, Steihaug H, Elvrum AG. Parental Coping, Representations, and Interactions with Their Infants at High Risk of Cerebral Palsy. J Clin Med. 2022 Dec 29;12(1):277. doi: 10.3390/jcm12010277. PMID 36615077